CLINICAL TRIAL: NCT07110818
Title: Improving Risk Prediction in Non-ischemic Cardiomyopathy (NICM): An Individualized Multimodality Approach Registry, Biobank and Imaging Data Repository
Brief Title: Non-ischemic Cardiomyopathy Registry, Biobank and Imaging Data Repository
Acronym: CaNICM
Status: Recruiting | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MP-33-2024-3373
Record Dates: First submitted 2025-06-03; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Non-ischemic Cardiomyopathy
Keywords: genetic; echocardiography; cardiac magnetic resonance imaging; biomarker; risk prediction model

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — DNA isolated from blood or saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main goal of CaNICM is to create a central database that includes a biobank and an imaging data repository for patients with non-ischemic cardiomyopathy (NICM), as well as for at-risk family members. This includes people who carry rare genetic variants linked to NICM but do not show symptoms, and first-degree relatives.

The specific goals of this database and biobank are to:

Enhance investigators' ability to predict the risk of heart rhythm disorders in patients with NICM.

Optimize the timing and approach for screening family members who may carry the disease - determining who to test, when, and how.

Find the best ways to treat family members early to prevent or slow the disease.

Future Phase - Phase 2 Goal:

4. Prospectively evaluate how well this risk prediction model works in real-life clinical settings, and compare it to the current approach, which is often based on a single risk factor.

DETAILED DESCRIPTION:
PATIENT ENROLLMENT:

Eligible patients will be included from collaborating centres. Patients will be contacted by the local investigator or a research coordinator. Willing individuals will be interviewed by the research coordinator and given information about biobank. The consent form will be reviewed and discussed with the coordinator. The investigators will also be available for any questions that the coordinator is unable to answer. Potential participants will have sufficient time to consider participating in CaNICM. Written informed consent will be obtained from eligible patients or legal guardians. Participants will be able to withdraw their participation at any time.

BASELINE DATA COLLECTION:

Clinical data will be collected from consented participants from the electronic medical report and a questionnaire. Images including CMR and Transthoracic echography (TTE) will be collected. ECG in the XML format will also be transferred. Blood samples will be collected for biobanking

Healthcare information will be coded in compliance with Tri Council Policy Statement criteria: direct identifiers will be removed and replaced with a unique study code (research CaNICM ID that does not use personal information such as the participant's health number, social insurance number or name. The coded data will be transferred into the clinical research database using a web-based electronic case report form (eCRF), using Redcap. The clinical research database will be hosted and managed at the Montreal Heart Institute Research center. The research ID uniquely identifying each subject eCRF within the database will be attributed by the research team but the master list of registry participants with their study identifiers will be kept separately from the clinical research database. This master list will be stored in an encrypted file within the research office of each site investigators under their supervision. Only the site investigators and their local research staff will have access to this list.

Baseline data collection and variables:

Baseline clinical data will be collected from consented participants from questionnaire. This includes demographic information and medical information such as the cardiac history, comorbidities, diagnostic test results, genetic testing results, family history and ethnicity, current and previous treatments. For patients who had had a CMR performed more than 2 years prior, baseline data will also be collected retrospectively at this time if available.

Based to contemporary practice (European society of Cardiology 2023 Cardiomyopathy guidelines8, EHRA/HRS/APHRS/LAHRS consensus on the state of genetic testing26 genetic testing will be recommended for probands and family members of families where the patient has a gene-causing variant.

BIOSPECIMEN COLLECTION:

Consented participants will undergo biosampling at enrollment for the primary purpose of DNA isolation and genetic studies. The preferred method is blood sampling using a standard venipuncture. Blood sampling allows for high quality DNA extraction as well as collection of plasma for potential future circulating biomarkers studies.

The CaNICM biobank will be directed by the Beaulieu-Saucier Pharmacogenomics Center (PGx; pharmacogenomics.ca/), operating under Good Laboratory/Clinical Practices (GLP/GCP) standards.

DNA isolation and long-term storage will be done at PGx, while long-term storage of plasma samples will be done at the MHI research center, in dedicated freezers located in a room with restricted access, under the supervision of Dr Julia Cadrin-Tourigny. All study samples will be stored for 50 years. Samples of subjects that withdraw their participation will be destroyed

IMAGING DATA TRANSFER:

For all consented participants, de-identified transthoracic echocardiography (TTE) and cardiac magnetic resonance (CMR) imaging data will be transferred to the Montreal Heart Institute imaging core-lab for central interpretation and long-term storage. At minimum, the following imaging studies are requested:

1. First available TTE
2. First available CMR, preferably with gadolinium injection
3. TTE closest to time of inclusion in the registry
4. CMR closest to time of inclusion in the registry
5. Last available TTE
6. Last available CMR, preferably with gadolinium injection

Digital Imaging and Communications in Medicine (DICOM) imaging data will be de-identified prior to transfer. De-identification will be performed at each site, by removing the patient's name and replacing the clinical identification number with the research CANICM ID. DICOM data will be stored using the Canadian Imaging network infrastructure (canadianimagingnetwork.org).

ECG data transfer:

For all consented participants, all de-identified ECG data in XML format will be transferred to the central database

Other:

Available relevant reports such as Holter reports and tracing, ICD implantation reports and intra-cardiac tracings will be transferred in the PDF format identified only by the study ID

PATIENT FOLLOW-UP:

Participants with a clinical diagnosis of NICM are expected to undergo yearly clinic visits, as per standard care. Participants without yearly clinic visits will be contacted by phone. Follow-up visits will assess for living status, functional class, medication as well as for arrhythmic, heart failure and thromboembolic events. A complete review of the medical record of the prior year will also be performed, including the transfer of medical notes from other hospitals where the participant has sought care if applicable. Follow-up data will be entered by the local investigator and/or research coordinator into an eCRF managed by the Montreal Heart Institute research center. De-identified documentation of clinical events including ECG, intracardiac tracing, clinical notes, imaging reports, and procedural reports will be uploaded to the database for centralized ad-hoc event adjudication.

De-identified DICOM images of TTE and CMR studies performed clinically during follow-up will be uploaded to the MHI imaging core-lab similarly as for baseline imaging studies.

For participants that will undergo biopsy, LVAD implantation or cardiac transplantation, surgical tissue samples will be collected using the Qiagen PAXgene tissue preservation system or equivalent, allowing for future somatic DNA, RNA and proteomic analyses. The samples will be stored at the MHI research center, under the supervision of Dr Julia Cadrin-Tourigny Upon enrollment, study subjects will be offered the option of providing an email contact information directly to the CaNICM study coordination center. This will allow the coordination center to directly contact participants to 1) provide study updates to participants, 2) obtain optional long-term follow-up data from participants, and 3) offer optional participation to future studies, including patient-reported outcome measures studies. At any time, participants can withdraw such contact information.

For family members, a follow-up every 3 years including an ECG, imaging (either TTE or CMR) and a Holter (PAC, NSVT) will be recommended.

ELIGIBILITY:
Inclusion Criteria:

1. LVEF <50% and/or
2. LVEF 50-55% with presence of clinically significant late gadolinium enhancement or LV dilatation and being carrier of a non ischemic cardiomyopathy causing gene (Pathogenic or likely pathogenic variant in a Clingen moderate or definite gene)

Exclusion Criteria:

* A significant other cause of decreased LVEF such as:

  1. Coronary artery stenosis (Significant lesion on proximal Left anterior descending or Left main, or ≥2 main branches with stenosis. Significant lesion is defined as >70% of any artery or >50% for the left main artery) or prior history of type 1 myocardial infarction
  2. Significant congenital heart disease requiring intervention
  3. Primary valvular disease including moderate to severe aortic stenosis and moderate to severe mitral stenosis, primary severe mitral regurgitation (secondary valvular disease such as mitral regurgitation/tricuspid regurgitation are not exclusion criteria)
  4. Other distinct entities: Amyloid heart disease, Chagas, Takotsubo, sarcoidosis, hemochromatosis related cardiomyopathy, HIV related cardiomyopathy are excluded
  5. Substances/therapies induced cardiomyopathy only if they are deemed to be the sole explanation for the cardiomyopathy (at the discretion of the enrolling cardiologist)
  6. Clear history of burned out hypertrophic cardiomyopathy
  7. Already had a transplantation at time of first CMR
  8. Refusal to provide informed consent

Additional remarks:

Patients aged > 70 years of age at first contact with a cardiologist regarding the cardiomyopathy will be limited to maximum 10% of the total enrolled patients by center.

Patients with risk factors (for example, chemotherapy, radiotherapy, alcohol…) for cardiomyopathy are not excluded unless they are deemed to completely account for the phenotype per the treating physician.

The inclusion is not restricted to adult patients and is planned to be extended to the pediatric population.

All included patients are recommended to have a CMR performed within 3 years of inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with NICM (non-schemic cardiomyopathy) as well as at-risk family members including unaffected carriers of rare genetic variants in genes causing NICM and first degree family members
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to first sustained ventricular arrhythmia | 5 years
  Spontaneous sustained VT
  ICD intervention (shock or antitachycardia pacing)
  Aborted sudden cardiac arrest (SCA)
  Sudden cardiac death (SCD)
Time to first life-threatening ventricular arrhythmia | 5 years
  defined as VT with a cycle length ≤ 240 ms (≥250 bpm)
Time to (aborted) sudden cardiac death in non-ICD carriers | 5 years
Atrial fibrillation and thromboembolic events: | 5 years
  Atrial fibrillation
  Stroke or systemic embolism

SECONDARY OUTCOMES:
Number of hospitalization or emergency visit for worsening heart failure | 5 years
Rate of end-Stage HF | 5 years
  Composite of heart transplant, mechanical cardiac support implantation, or cardiovascular death.
Number of clinical HF | 5 years
  Composite of hospitalization or emergency room visit for HF (admission primarily for HF and worsening HF requiring intensification of HF treatment), new prescription of loop diuretic or LVEF decline to <40% with change ≥ 10% from baseline (TTE or CMR).

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No